CLINICAL TRIAL: NCT02418143
Title: A Post Market Observational Study to Obtain Additional Information on the Use of CorMatrix® CanGaroo ECM® Envelope
Brief Title: A Study to Obtain Additional Information on the Use of CorMatrix® CanGaroo ECM® Envelope
Acronym: JUMP
Status: Withdrawn | Type: Observational
Sponsor: Elutia Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 15-PR-1169
Record Dates: First submitted 2015-04-09; First posted 2015-04-16 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Implantable electronic device placement: CorMatrix CanGaroo ECM envelope for an implantable electronic device placement following a battery change out or upgrade.
  Interventions: Device: CorMatrix CanGaroo ECM Envelope

INTERVENTIONS:
Device: CorMatrix CanGaroo ECM Envelope — Subjects who have received CorMatrix CanGaroo ECM Envelope for an implantable electronic device placement following a battery change or upgrade.

SUMMARY:
Actively gather additional information on the use of CorMatrix CanGaroo ECM Envelope in a post market observational study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who has received the CorMatrix CanGaroo ECM Envelope for an implantable electronic device following battery change out or upgrade.
2. Signed Informed Consent

Exclusion Criteria:

1. Known sensitivities to porcine material.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of any subject who has received the CorMatrix CanGaroo ECM Envelope for an implantable electronic device placement following a battery change out or upgrade.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Device Related Adverse Events | 1 day post-operative follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Director, Clinical Development, Study Director — Aziyo Biologics